CLINICAL TRIAL: NCT04411758
Title: Propolis as a New Strategy in Modulating Inflammation in Patients With Chronic Kidney Disease.
Brief Title: Propolis for Patients With Chronic Kidney Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Denise Mafra8
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Chronic Kidney Diseases; Inflammation
Keywords: chronic kidney disease; non-dialysis; propolis; inflammation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation | interventions — Propolis

STUDY DESIGN:
Intervention Model Description: In this clinical trial, participants with CKD undergoing hemodialysis or peritoneal dialysis will be instructed to use 4 capsules of 500mg/day containing concentrated and standardized dry green propolis extract (EPP-AF®) for 2 months or placebo (4 capsules of 500mg/day of magnesium stearate, silicon dioxide and microcrystalline cellulose) for two months, and then the groups will be crossed and will receive the same amount of propolis as the first group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Patients will receive 4 capsules (400mg/day) containing magnesium stearate, silicon dioxide and microcrystalline cellulose for 2 months
  Interventions: Dietary Supplement: Placebo
- Propolis Group (Experimental): Patients will receive 4 capsules (400mg/day) containing dry EPP-AF® green propolis extract for 2 months
  Interventions: Dietary Supplement: Propolis

INTERVENTIONS:
Dietary Supplement: Propolis — Four capsules (400mg/day) containing dry EPP-AF® green propolis extract for 2 months and after washout, more two months crossover
  Arms: Propolis Group
Dietary Supplement: Placebo — Four capsules (400mg/day) containing magnesium stearate, silicon dioxide and microcrystalline cellulose for 2 months and after washout, more two months crossover
  Arms: Placebo Group

SUMMARY:
To evaluate the effects of propolis extract on inflammation in participants with chronic kidney disease.

Specific objectives

To assess before and after the intervention period:

* The expression of transcription factors (nuclear factor-kB), antioxidant enzymes (heme-oxygenase-1), inflammasome receptor, peroxisome proliferator-activated receptor-γ, as well as the levels of inflammatory cytokines (IL-6, Tumor nuclear factor-α, C-reactive protein, interleukin 1) and E-selectin adhesion molecules;
* The levels of protein expression of inflammatory markers and antioxidant enzymes;
* The profile of the intestinal microbiota of stool samples from the research participants;
* Plasma levels of substances reactive to thiobarbituric acid and oxidized low density lipoprotein as a marker of oxidative stress;
* Routine and anthropometric laboratory variables, indicative of the metabolic profile of the research participants;
* Assess blood pressure, 6-minute walk test, recovery heart rate and chair lift test to assess the functional capacity of the research participants;
* Assess atherogenic risk;
* Food intake and nutritional status; Compare data between the intervention and control groups.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) has chronic systemic inflammation as an important component of multifactorial origin, a factor related to both the progression and outcomes of CKD, being involved in all causes of mortality in these patients, such as cardiovascular disease. In this context, some nutritional strategies have been proposed as an adjuvant therapeutic alternative to modulate inflammation, starting from the consolidated knowledge of the role of nutrients and bioactive compounds on the expression of genes related to inflammation and oxidative stress, factors that feed on each other. In view of this scenario, propolis, a substance made up of a combination of several chemical components with broad potential biological activity, appears as a promising alternative to modulate inflammation in patients with CKD. However, clinical evidence to assess the effects of propolis in patients with CKD is scarce, and there are no studies that have investigated its effects on gene expression and markers related to inflammation in these patients. Thus, the present project proposes a longitudinal study of the clinical trial type that aims to evaluate the effects of propolis alcoholic extract on transcription factors and inflammatory markers in patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

• Aged 18 years or older

- with fistula arteriovenous

Exclusion Criteria:

* Patients pregnant
* Smokers
* Using antibiotics in the last three months
* Using antioxidant supplements as antioxidant vitamins, probiotic, prebiotic, symbiotic and antibiotics in the last three months
* Clinical diagnosis of infectious diseases
* Clinical diagnosis of Cancer
* Clinical diagnosis of AIDS - for PD patients - no peritonitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in cytokines plasma levels measured by ELISA after supplementation with propolis. | 4 months
  IL-6, Tumor necrosis factor (TNF)
Change the expression of transcription factors (nuclear factor-kB), antioxidant enzymes (heme-oxygenase-1), inflammasome, peroxisome proliferator-activated receptor-γ | 4 months
  nuclear factor (NF)-kappa B
Change the profile of the intestinal microbiota of stool samples | 4 months
  uremic toxins

CONTACTS AND LOCATIONS:
Overall Officials: Denise Mafra, phd, Principal Investigator — Universidade Federal Fluminense
Locations (1):
- Denise Mafra, Niterói, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fonseca L, Ribeiro M, Schultz J, Borges NA, Cardozo L, Leal VO, Ribeiro-Alves M, Paiva BR, Leite PEC, Sanz CL, Kussi F, Nakao LS, Rosado A, Stenvinkel P, Mafra D. Effects of Propolis Supplementation on Gut Microbiota and Uremic Toxin Profiles of Patients Undergoing Hemodialysis. Toxins (Basel). 2024 Sep 25;16(10):416. doi: 10.3390/toxins16100416. PMID 39453192
- [Derived] Baptista BG, Fanton S, Ribeiro M, Cardozo LF, Regis B, Alvarenga L, Ribeiro-Alves M, Berretta AA, Shiels PG, Mafra D. The effect of Brazilian Green Propolis extract on inflammation in patients with chronic kidney disease on peritoneal dialysis: A randomised double-blind controlled clinical trial. Phytomedicine. 2023 Jun;114:154731. doi: 10.1016/j.phymed.2023.154731. Epub 2023 Mar 1. PMID 36934668
- [Derived] Chermut TR, Fonseca L, Figueiredo N, de Oliveira Leal V, Borges NA, Cardozo LF, Correa Leite PE, Alvarenga L, Regis B, Delgado A, Berretta AA, Ribeiro-Alves M, Mafra D. Effects of propolis on inflammation markers in patients undergoing hemodialysis: A randomized, double-blind controlled clinical trial. Complement Ther Clin Pract. 2023 May;51:101732. doi: 10.1016/j.ctcp.2023.101732. Epub 2023 Jan 26. PMID 36708650